CLINICAL TRIAL: NCT06733805
Title: Impact Evaluation of the Therapeutic Initiative's Type 2 Diabetes in Older Adults Portrait and Therapeutics Letter
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Health, British Columbia (Other Government)
Responsible Party: Principal Investigator, Colin Dormuth, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: H24-01347
Record Dates: First submitted 2024-11-19; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Clinical Audit; Quality Improvement; T2DM (Type 2 Diabetes Mellitus)
Keywords: Randomized controlled trial; Type 2 Diabetes in older adults; Quality improvement; Prescribing feedback
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The investigators randomized actively practicing family physicians and nurse practitioners into two groups, n = 3,407 in each group. They then looked at who was registered for Portrait Online at the time of generating the early portrait data, and there were n=259 in Group 1, and n=256 in Group 2 for a total of 515 individuals.
  Group 1 received the intervention materials on January 15, 2024, while Group 2 received nothing (thus serving as the control group). Group 2 received the intervention materials nine months later, on October 15, 2024.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Early Portrait + Letter (Experimental): This group received the prescribing portrait and therapeutics letter on January 15, 2024. The materials were uploaded to the Portrait Online interface on this date, and recipients were sent an email notifying them of the new material available.
  Interventions: Behavioral: Portrait + Therapeutics Letter
- Group 2 - Delayed Control (Experimental): This group received the prescribing portrait and therapeutics letter on October 15, 2024 (9 months after Group 1 received the materials). The materials were uploaded to the Portrait Online interface on this date, and recipients were sent an email notifying them of the new material available.
  Interventions: Behavioral: Portrait + Therapeutics Letter

INTERVENTIONS:
Behavioral: Portrait + Therapeutics Letter — In the context of audit and feedback interventions, Portrait is a document produced by the physician organization Therapeutics Initiative that provides personalized prescribing feedback for BC clinicians. Portraits are used as a practice resource tool for reflection on prescribing patterns. Each Portrait topic provides data of individual prescriber's prescribing practice, benchmarks or targets, a succinct review of the best-available evidence on the topic, and recommendations for future action.
  The Therapeutics Letter is a standalone publication that details identified problematic therapeutic issues in a brief, simple and practical manner. Therapeutics letters include a systematic literature review on a clinical topic, and provide reference for the data presented in the Portraits.

SUMMARY:
The goal of this randomized trial is to learn if educational materials and personalized prescribing portraits change how clinicians in British Columbia (BC), Canada treat older adults with type 2 diabetes (T2DM). The main question the investigators aim to answer is:

• Did a personalized prescribing portrait and therapeutics letter lead to a change in the number of older adults prescribed sulfonylureas or insulin when they have glycated hemoglobin (A1C) levels below 7%, compared to usual care.

Study participants are nurse practitioners and family physicians actively practicing in BC, Canada. Participants registered on the project website, Portrait Online, to receive their digital prescribing portraits. Participants were randomized to either receive educational materials in the Early Group or in the Delayed Group. Using administrative health data, the prescribing of those in the Early Group will be compared to those in the Delayed Group to see if the materials influenced their prescribing.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) is common in older adults (65 years and older). Older adults are more likely to experience negative effects of medications used to treat T2DM, especially low blood sugar. Low blood sugar is dangerous for older adults and can lead to a higher risk of hospitalization. Medications such as insulins or sulfonylureas carry the highest risk of low blood sugar. Available evidence suggests that using insulin or sulfonylureas to treat T2DM to aggressive targets (glycated hemoglobin [A1C] less than 7%) does more harm than good. Therefore, insulin and sulfonylureas are not recommended for older adults with A1C less than 7%. Unfortunately, insulin and sulfonylurea use remains common among older adults living with T2DM.

Audit and feedback is an approach where individual prescribers receive feedback on their own prescribing (and may be compared to a benchmark) with the aim of improving their prescribing. This may be accompanied by education on how and why to improve. The investigators' research group does regular work in this area through the Portrait program, which aims to improve prescribing by providing audit and feedback and education to prescribers in British Columbia (BC), Canada.

This study is a randomized trial testing the effectiveness of personalized prescribing Portraits and Therapeutics Letters on prescribing of sulfonylureas and insulins for older patients with T2DM in the primary care setting in the Canadian province of BC.

6,814 active BC clinicians (family physicians and nurse practitioners) were randomly divided into 2 groups (n =3,407 in each group). At the time the Portraits were generated, there were 515 people registered for Portrait Online, the secure website through which clinicians are able to receive their confidential Portraits (Group 1, n = 259; Group 2, n = 256).

On January 15, 2024 Group 1 clinicians were notified by email that their prescribing Portraits and Therapeutics Letter were available for viewing in their Portrait Online accounts. Nine months later, on October 15, 2024, clinicians in Group 2 received this same notification and access to the same materials. The analysis will assess whether the materials led Group 1 clinicians to change how they prescribe sulfonylureas and insulins to older people with T2DM.

The analysis will include:

* Baseline characteristics of physicians and patients by study group
* Trends in monthly prescribing for all of BC of sulfonylureas and insulins from 1 year prior to release of the materials to the end of the study (January 15, 2023 to January 15, 2025). This will illustrate background trends in prescribing patterns.
* Difference in change from baseline for mean number of patients with A1C < 7% taking a sulfonylurea or insulin between Group 1 and Group 2.
* Proportion of patients with an A1C ≤ 7% who are newly started on a sulfonylurea or insulin by Group 1 prescribers compared to the proportion in the matched control group (Group 2).

Analysis will be conducted using secondary data from administrative databases from the BC Ministry of Health (under an Information Sharing Agreement). The data are patient level and include anonymized information about demographics, health costs, physician billing codes, prescriptions, outpatient records, and hospitalizations. The data do not include personally identifiable patient information.

ELIGIBILITY:
Inclusion Criteria:

* Registered with the College of Physicians and Surgeons of BC or BC College of Nurses and Midwives as a nurse practitioner.
* For physicians: defined as a General Practitioner or Family Physician - Emergency Medicine according to the BC Ministry of Health's Medical Services Plan with a license status of private practice, temporary license, salaried, or post graduate.
* Had ≥100 patients with prescriptions filled at a community pharmacy in 2022.
* Registered for Portrait Online (the program's secure website).

Exclusion Criteria:

* Not registered with the College of Physicians and Surgeons of BC or BC College of Nurses and Midwives as a nurse practitioner.
* Physicians who were not classified as a General Practitioner or Family Practice - Emergency Medicine according to the BC Ministry of Health's Medical Services Plan with a license status of private practice, temporary license, salaried, or post graduate.
* Had fewer than 100 patients with prescriptions filled at a community pharmacy in 2022.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 515 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Difference in change from baseline for mean number of patients with A1C < 7% taking a study drug between Group 1 and Group 2 | 9 months
  The primary outcome is the difference in the change from baseline in the mean number of patients with A1C ≤ 7% taking a sulfonylurea or insulin at 9-months after the early release of the Portrait and Therapeutics Letter (intention-to-treat analysis). The investigators will use a 2-sample t-test, with an alpha of 0.05 to test for statistical significance.

SECONDARY OUTCOMES:
Difference in change from baseline for mean number of patients with A1C < 7% taking a study drug between Group 1 who opened the Portrait and Group 2 | 9 months
  The secondary outcome is the difference in the change from baseline in the mean number of patients with A1C ≤ 7% taking a sulfonylurea or insulin at 9-months after the early release of the Portrait for prescribers who opened the Portrait (per-protocol analysis). The investigators will use a 2-sample t-test, with an alpha of 0.05 to test for statistical significance.

OTHER OUTCOMES:
Change from baseline in new starts of a study drug for patients with an A1C ≤ 7% between Group 1 who opened the Portrait and Group 2 | Up to 9 months
  The tertiary outcome is new starts of a sulfonylurea or insulin for patients with an A1C ≤ 7% from baseline to 9-months for prescribers who opened their Portrait (per-protocol-analysis). For this analysis, baseline will be the date when the prescriber opened their Portrait. The comparator will be matched to practitioners from the delay arm who are registered for Portrait Online (matched on age (+/- 5 years), sex, urban/rural practice location, nurse practitioner/family physician) in up-to a 3:1 ratio. The investigators will calculate a relative risk and 95% CI and adjust for clustering using generalized estimating equations.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Dormuth, ScD, Principal Investigator — University of British Columbia
Locations (1):
- Therapeutics Initiative - Dept of Anesthesiology, Pharmacology & Therapeutics, Faculty of Medicine, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
This study's data access does not permit sharing of individual participant data. Access to administrative data can be requested through the BC Ministry of Health.